CLINICAL TRIAL: NCT04078243
Title: Feasibility of Novel Clinical Trial Infrastructure, Design and Technology for Early Phase Studies in Patients With Pulmonary Hypertension.
Brief Title: Feasibility of Novel Clinical Trial Infrastructure, Design and Technology for Early Phase Studies in Patients With Pulmonary Hypertension (FIT-PH)
Acronym: FIT-PH
Status: Recruiting | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH20422
Record Dates: First submitted 2019-08-21; First posted 2019-09-06 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CardioMEMS HF System: Eligible patients will be recruited and will attend for the implantation in line with standard of care procedures. The patient's details will be uploaded to the CardioMEMS HF system, enabling remote monitoring of their heart failure device. The patient will also be given a Fitbit activity monitor and set up with an account that is accessible to patient and physician to allowing activity to be monitored. The research team will be able to continuously monitor data remotely from the CardioMEMS HF system and Fitbit platform.
  Interventions: Device: CardioMEMS HF System

INTERVENTIONS:
Device: CardioMEMS HF System — The CardioMEMS HF System is the first and only FDA-approved wireless heart failure monitor. The system is a safe, reliable way to help your patients manage their heart failure.

SUMMARY:
Prospective, open-label, observational study to evaluate the safety and feasibility of using pulmonary artery pressure (PAP) monitors and wearable activity monitors in patients with pulmonary hypertension (PH).

DETAILED DESCRIPTION:
This is a prospective, open-label, observational study, to evaluate the safety and feasibility of using pulmonary artery pressure monitors and wearable activity monitors in patients with pulmonary hypertension. We plan to correlate data from the PAP monitors with data from wearable activity monitors and review how often patients require ad hoc visits / medication changes as well as review the optimum dose of drug achieved / patient QoL / risk stratification and patient outcomes / mortality.

Suitable patients, with a confirmed diagnosis of PH on RHC, will be recruited from outpatient clinic or day-case and ward admissions by physicians or the research team. A face to face or telephone conversation will occur to discuss the study in detail and if the patient is willing they will be given / sent a patient information sheet (PIS) and be invited to attend a screening visit. If eligibility criteria are met, patients will complete a consent form and have their medical history reviewed including but not limited to past medical history, medication review, allergies and review of any hospital admissions in the previous 12 months. A clinical examination with observations including, but not limited to blood pressure, heart rate, oxygen saturations, respiratory rate, temperature, weight, height, body mass index (BMI) and assessment of NYHA class will be undertaken. Patients will be asked to perform a baseline six minute walk test, complete a quality of life questionnaire (EMPHASIS-10), 12-Lead ECG and baseline, clinically-indicated blood testing (including but not limited to FBC,UE,LFT, clotting screen, NT-Pro BNP) and imaging performed in clinical practise (TTE or cardiac MRI) will be reviewed. Eligible subjects will be scheduled for the Implant procedure. Subjects on anticoagulation therapy (e.g. warfarin) may be instructed by the Investigator to discontinue use 2 days prior to pressure sensor placement and may be bridged with low molecular weight heparin if required according to local trust standard of care bridging protocol.

If eligible, patients will then attend for their implantation visit and at this point undergo a RHC and a CardioMEMSTM sensor implant in the catheter laboratory. Baseline readings will be taken from the pressure monitor (including systolic, mean and diastolic PAP and cardiac output) and calibrated with readings taken at RHC. The patient's details will be uploaded to the CardioMEMSTM HF system, enabling remote monitoring of their heart failure device. Time will be spent educating and familiarising the patient with the home monitor system and contact details given in case any issues arise on discharge. Patients will be advised to submit one reading per day, preferably at the same time of day and in the same position i.e. lying down flat or at 45 degrees etc. Patients will be asked to monitor their symptom burden and to share this with the investigators.

The patient will also be given a Fitbit activity monitor and set up with an account that is accessible to patient and physician to allowing activity to be monitored. The research team will be able to continuously monitor data remotely from the CardioMEMSTM HF system and Fitbit platform.

Patients will attend for follow-up visits at 30 days and 1 year and will have their history reviewed and clinical examination and observations reassessed. At this point a repeat 6MWT, emPHasis-10 questionnaire, NYHA functional class and 12 Lead ECG will be undertaken as well as bloods testing and imaging as clinically indicated. Readings from the CardioMEMSTM HF system and Fitbit platform will also be reviewed and compared to the patients symptom diary.

In between visits patients will be contacted by telephone and invited for unscheduled visits if clinically indicated. Any clinically significant data or medication changes will be discussed or fed back to the clinical PH team in charge of the patients routine care as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pulmonary hypertension (Group I,II,III and IV)
* Age 18 years
* Estimated glomerular filtration rate (eGFR) > 25
* Body mass index (BMI) < 35 (or equivalent)
* Pulmonary artery (PA) branch 7mm
* Negative pregnancy test (If female of childbearing age)
* Written, informed consent completed
* Willingness of the patient to comply

Exclusion Criteria:

* Group IV PH
* Active infection
* Pulmonary embolus (PE) or deep vein thrombosis (DVT)
* Major cardiovascular event within past 2 months
* Cardiac resynchronisation therapy (CRT) device within past 3 months
* Mechanical right heart valve
* Known coagulation disorder
* Known hypersensitivity to aspirin or clopidogrel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of PH at right heart catheterisation (RHC) and New York Heart Association (NYHA) class III, prior admission for treatment of heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2028-01-06 (Estimated); Study Completion 2028-09-06 (Estimated)

PRIMARY OUTCOMES:
Activity Monitors | Through study completion - 30/03/2024
  To test the safety and feasibility of pressure monitoring and wearable activity monitors in patients with PH.

SECONDARY OUTCOMES:
Pulmonary Artery Pressure | Through study completion - 30/03/2024
  To correlate Pulmonary Artery Pressure changes with outcome and activity data.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galie N, McLaughlin VV, Rubin LJ, Simonneau G. An overview of the 6th World Symposium on Pulmonary Hypertension. Eur Respir J. 2019 Jan 24;53(1):1802148. doi: 10.1183/13993003.02148-2018. Print 2019 Jan. PMID 30552088
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113
- [Background] Koehler F, Koehler K, Deckwart O, Prescher S, Wegscheider K, Kirwan BA, Winkler S, Vettorazzi E, Bruch L, Oeff M, Zugck C, Doerr G, Naegele H, Stork S, Butter C, Sechtem U, Angermann C, Gola G, Prondzinsky R, Edelmann F, Spethmann S, Schellong SM, Schulze PC, Bauersachs J, Wellge B, Schoebel C, Tajsic M, Dreger H, Anker SD, Stangl K. Efficacy of telemedical interventional management in patients with heart failure (TIM-HF2): a randomised, controlled, parallel-group, unmasked trial. Lancet. 2018 Sep 22;392(10152):1047-1057. doi: 10.1016/S0140-6736(18)31880-4. Epub 2018 Aug 25. PMID 30153985
- [Background] Adamson PB. Pathophysiology of the transition from chronic compensated and acute decompensated heart failure: new insights from continuous monitoring devices. Curr Heart Fail Rep. 2009 Dec;6(4):287-92. doi: 10.1007/s11897-009-0039-z. PMID 19948098
- [Background] Adamson PB, Magalski A, Braunschweig F, Bohm M, Reynolds D, Steinhaus D, Luby A, Linde C, Ryden L, Cremers B, Takle T, Bennett T. Ongoing right ventricular hemodynamics in heart failure: clinical value of measurements derived from an implantable monitoring system. J Am Coll Cardiol. 2003 Feb 19;41(4):565-71. doi: 10.1016/s0735-1097(02)02896-6. PMID 12598066
- [Background] Zile MR, Bennett TD, St John Sutton M, Cho YK, Adamson PB, Aaron MF, Aranda JM Jr, Abraham WT, Smart FW, Stevenson LW, Kueffer FJ, Bourge RC. Transition from chronic compensated to acute decompensated heart failure: pathophysiological insights obtained from continuous monitoring of intracardiac pressures. Circulation. 2008 Sep 30;118(14):1433-41. doi: 10.1161/CIRCULATIONAHA.108.783910. Epub 2008 Sep 15. PMID 18794390
- [Background] Adamson PB, Abraham WT, Aaron M, Aranda JM Jr, Bourge RC, Smith A, Stevenson LW, Bauman JG, Yadav JS. CHAMPION trial rationale and design: the long-term safety and clinical efficacy of a wireless pulmonary artery pressure monitoring system. J Card Fail. 2011 Jan;17(1):3-10. doi: 10.1016/j.cardfail.2010.08.002. PMID 21187258
- [Background] Givertz MM, Stevenson LW, Costanzo MR, Bourge RC, Bauman JG, Ginn G, Abraham WT; CHAMPION Trial Investigators. Pulmonary Artery Pressure-Guided Management of Patients With Heart Failure and Reduced Ejection Fraction. J Am Coll Cardiol. 2017 Oct 10;70(15):1875-1886. doi: 10.1016/j.jacc.2017.08.010. PMID 28982501
- [Background] Abraham WT, Adamson PB, Hasan A, Bourge RC, Pamboukian SV, Aaron MF, Raval NY. Safety and accuracy of a wireless pulmonary artery pressure monitoring system in patients with heart failure. Am Heart J. 2011 Mar;161(3):558-66. doi: 10.1016/j.ahj.2010.10.041. Epub 2011 Jan 31. PMID 21392612
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Raeside DA, Chalmers G, Clelland J, Madhok R, Peacock AJ. Pulmonary artery pressure variation in patients with connective tissue disease: 24 hour ambulatory pulmonary artery pressure monitoring. Thorax. 1998 Oct;53(10):857-62. doi: 10.1136/thx.53.10.857. PMID 10193372
- [Background] Redfield MM, Anstrom KJ, Levine JA, Koepp GA, Borlaug BA, Chen HH, LeWinter MM, Joseph SM, Shah SJ, Semigran MJ, Felker GM, Cole RT, Reeves GR, Tedford RJ, Tang WH, McNulty SE, Velazquez EJ, Shah MR, Braunwald E; NHLBI Heart Failure Clinical Research Network. Isosorbide Mononitrate in Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2015 Dec 10;373(24):2314-24. doi: 10.1056/NEJMoa1510774. Epub 2015 Nov 8. PMID 26549714
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Yorke J, Corris P, Gaine S, Gibbs JS, Kiely DG, Harries C, Pollock V, Armstrong I. emPHasis-10: development of a health-related quality of life measure in pulmonary hypertension. Eur Respir J. 2014 Apr;43(4):1106-13. doi: 10.1183/09031936.00127113. Epub 2013 Nov 14. PMID 24232702